CLINICAL TRIAL: NCT04457206
Title: Evaluating the Effectiveness of the Collaborative Community Clinic for Persons With Spinal Cord Injury and Disease
Brief Title: Effectiveness of the Collaborative Community Clinic for Persons With Spinal Cord Injury and Disease
Acronym: SCI/D
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Carla Walker, Principal Investigator, Washington University School of Medicine
Other Study IDs: 202001182
Record Dates: First submitted 2020-06-24; First posted 2020-07-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: SCI Group and one-on-one services through student led occupational therapy clinic — The Collaborative Community Clinic (CCC) students collaborate with Dr. Walker to conduct the spinal cord injury/disease (SCI/D) Health and Participation Program, which consists of a combination of groups and one-on-one OT sessions serving persons with spinal cord injury and disease who are un- or under-insured. The program includes a pre-assessment session, four groups, optional individual sessions and a post-survey. Group topics include bowel/bladder management, community mobility, advocacy, transportation, promoting intimacy, adaptive parenting and finding resources. Students are involved in recruiting participants, co-leading group sessions, treatment planning and implementation for individual sessions, and development of topic-specific materials.

SUMMARY:
The investigator is evaluating data stored on the Collaborative Community Clinic data repository (IRB #201811032). Researchers seek to evaluate the effectiveness of the Collaborative Community Clinic (CCC), an occupational therapy student experiential learning clinic for uninsured or under-insured people with spinal cord injury and disease (SCI/D), using participants' initial and follow-up assessment batteries.

DETAILED DESCRIPTION:
All data reviewed will be pulled from the Collaborative Community Clinic (CCC) data repository according to the data manual and procedures. A separate IRB was approved to review outcomes from participants in the CCC to evaluate the effectiveness of the clinic. All participants participated in an informed consent process to provide the option to have their data stored in a data repository for aggregate review. If any participate chooses not to have their data stored, it will not be stored or outcomes reviewed. However, participants are still provided services through the CCC. Researchers anticipate up to 200 participants participating in the registry over five years. All data will be data checked by a member of the research team to limit errors and identification of missing data recorded. Statistical analysis methods are to be determined upon completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age; diagnosis of spinal cord injury or disease, un-insured or under-insured for occupational therapy services

Exclusion Criteria:

* under 18 years of age, lack of SCI/D diagnosis, full insurance coverage for OT services (ie. Medicare or Private Insurance)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persons participating in the Collaborative Community Clinic are 18 years of age or older, have the diagnosis of spinal cord injury or disease and are un-insured or under-insured for occupational therapy services. For example, they may have Medicaid coverage, but no therapy visits allowed. Or, they may be waiting on Medicare eligibility to kick in following injury, which usually takes approximately two years. Persons may be referred following discharge from the local rehabilitation center, be referred from other community agencies, or self-referred.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2030-01-29 (Estimated); Study Completion 2030-01-29 (Estimated)

PRIMARY OUTCOMES:
General Self-Efficacy Scale | pre-assessment before participation in the CCC and post-assessment following completion (approximately 12 weeks)
  When completing the General Self-Efficacy Scale, clients rate a series of statements intended to measure feelings of self-efficacy such as "I can always manage to solve difficult problems if I try hard enough" on a scale of 1 (not at all true) to 4 (exactly true).It evaluates change in ability to self-manage health before and after participation in the Collaborative Community Clinic (CCC).
The Canadian Occupational Performance Measure (COPM) | pre-assessment before participation in the CCC and post-assessment upon completion of CCC participation (approximately 12 weeks)
  The COPM measures perceived change in occupational performance. Each scale rated on a scale of 1 (low) to 10 (high). It is an evidence-based outcome measure designed to capture a participant's change in self-perception of performance in everyday living, over time before participation in the CCC and upon completion. The COPM has a broad focus on occupational performance in all areas of life, including self-care, leisure, and productivity, considering circumstances across the lifespan.

SECONDARY OUTCOMES:
Promis 29 Global Health Measure | pre-assessment prior to participation in the CCC and post-assessment upone completion of CCC participation (approximately 12 weeks)
  The PROMIS-29 is a collection of four-item individual short forms assessing change in seven different domains: anxiety, depression, fatigue, pain interference, physical function, sleep disturbance, and ability to participate in social roles and activities, as well as a single pain intensity item. Individuals respond to the four items in each domain using a five-point Likert scale (5: without any difficulty, 1: unable to do). *T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points.
Community Participation Index (CPI): | pre-assessment prior to participation in the CCC and post-assessment upon completion of the CCC participation (approximately 12 weeks)
  The CPI is a valid and reliable assessment of change in involvement in life situations and individual control over participation. For each item, respondents rate frequency (in days, hours, or times per week, depending on the activity), whether it is important (yes/no), and to what extent they do the item (too much, enough, or not enough). The measure is used as a categorical variable using validated scores. Participation will be assessed at baseline and upon completion of the group and individual visits. A percentage satisfaction with community participation in achieved by totaling the number of items important to them, that they are doing enough of divided by the total number of activities that were listed as important to them and multiplying by 100. So, if 20 activities were important and 6 were being completed enough, they would have a 30% satisifaction rate (6/20 x100)
PROMIS Item Bank v1.0 - Emotional Distress - Depression-Short Form 8a | pre-assessment prior to participation in the CCC and post-assessment upon completion of participation in the CCC (approximately 12 weeks)
  short form depression scale - self-report - Change in scores with participation in the CCC. *T-Scores are used to interpret severity of depression by the following: 55 and under indicating slight to none, 55-59.9 mild, 60-69.9 moderate, and 70+ indicating severe.
Promis Item Bank v1.0 - Applied Cognition-Abilities Short Form 8a | pre-assessment prior to participation in the CCC and post-assessment upon completion of participation in the CCC (approximately 12 weeks)
  short self-report of changes in cognition. *T-Score distributions are standardized such that a 50 represents the average (mean) for the US general population, and the standard deviation around that mean is 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Carla W Walker, OTD, Principal Investigator — Washington University Program in Occupational Therapy
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share participant data with other researchers at this time.

REFERENCES:
- [Background] Garber SL, Rintala DH, Hart KA, Fuhrer MJ. Pressure ulcer risk in spinal cord injury: predictors of ulcer status over 3 years. Arch Phys Med Rehabil. 2000 Apr;81(4):465-71. doi: 10.1053/mr.2000.3889. PMID 10768537
- [Background] Gray DB, Hollingsworth HH, Stark SL, Morgan KA. Participation survey/mobility: psychometric properties of a measure of participation for people with mobility impairments and limitations. Arch Phys Med Rehabil. 2006 Feb;87(2):189-97. doi: 10.1016/j.apmr.2005.09.014. PMID 16442971
- [Background] Miller LC, Gottlieb M, Morgan KA, Gray DB. Interviews with employed people with mobility impairments and limitations: environmental supports impacting work acquisition and satisfaction. Work. 2014;48(3):361-72. doi: 10.3233/WOR-131784. PMID 24284677
- [Result] Craig A, Tran Y, Middleton J. Psychological morbidity and spinal cord injury: a systematic review. Spinal Cord. 2009 Feb;47(2):108-14. doi: 10.1038/sc.2008.115. Epub 2008 Sep 9. PMID 18779835
- See also: paralyzed veterans of america website — https://www.pva.org/spinal-cord-injury-information